CLINICAL TRIAL: NCT01376856
Title: Characteristics of Mediastinal Lymph Node With False Positive FDG PET/CT Results in Lung Cancer Staging : Relation With TB and Latent TB Infection
Status: Terminated | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0196
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: mediastinal lymph node with false positive FDG PET/CT results in lung cancer staging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood for perfoming Quantiferon-TB Gold in tube assay
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET/CT and surgical biopsy group: person who performed PET/CT and surgical biopsy of mediastinal lymph node for diagnosis of primary lung cancer of metastatic lung cancer

SUMMARY:
The purpose of this study is to analyze pathologic and radiologic characteristics of mediastinal lymph nodes with false positive FDG PET/CT results in lung cancer staging and assess relationship between false positive mediastinal lymph node and TB/latent TB.

ELIGIBILITY:
Inclusion Criteria:

* age 20-75, men and women
* person who performed PET/CT and surgical biopsy of mediastinal lymph node for diagnosis of primary lung cancer of metastatic lung cancer

Exclusion Criteria:

* age < 20
* person who don't agree with enrollment
* illiterate
* person who is diagnosed as active tuberculosis now
* person who has history of hypersensitivity on PPD (tuberculin purified protein derivative)
* pregnant woman
* person who is treated as active tuberculosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: person who performed PET/CT and surgical biposy of mediastinal lymph node for diagnosis of primary lung cancer of metastatic lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
false positive rate of Mediastinal Lymph Node | 3months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea